CLINICAL TRIAL: NCT00880815
Title: Fludarabine, Bendamustine, and Rituximab (FBR) Non-Myeloablative Allogeneic Conditioning for Patients With Lymphoid Malignancies
Brief Title: Fludarabine, Bendamustine, and Rituximab in Treating Participants With Lymphoid Cancers Undergoing Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0246; NCI-2018-01844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0246 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: CD20 Positive; Chronic Lymphocytic Leukemia; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell | interventions — Antilymphocyte Serum; thymoglobulin; Bendamustine Hydrochloride; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Methotrexate; merphos; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, stem cell transplant, rituximab) (Experimental): Participants receive rituximab IV over 5-7 hours on days -13 and -6, fludarabine IV over 1 hour and bendamustine IV over 1 hour on days -5 to -3, and tacrolimus IV starting on day -2 and PO after hospital discharge for 6 to 8 months. Participants with MUD receive thymoglobulin on days -2 and -1. Participants undergo allogenic stem cell transplant over 30-45 minutes on day 0. Participants receive rituximab IV over 5-7 hours on days 1 and 8 and methotrexate IV over 30 minutes on days 1, 3, and 6. Participants with MUD also receive methotrexate IV on day 11. Participants receive G-CSF SC once daily starting on day 7 until white blood cell counts recover.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Bendamustine; Biological: Filgrastim; Drug: Fludarabine; Drug: Methotrexate; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Biological: Filgrastim — Given IV
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase I trial studies the best dose and how well bendamustine works with standard chemotherapy (fludarabine, rituximab) in treating participants with lymphoid cancers undergoing stem cell transplant. Drugs used in chemotherapy, such as fludarabine, bendamustine, and rituximab, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a stem cell transplant helps stop the growth of cancer cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the participant, they may help the participant's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes, the transplanted cells from a donor can make an immune response against the body's normal cells called graft versus host disease. Giving rituximab and methotrexate after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine engraftment and dose limiting toxicity (DLT) of bendamustine in patients with lymphoid malignancies undergoing non-myeloablative allogeneic hematopoietic transplantation.

SECONDARY OBJECTIVES:

I. To monitor the risk of graft-versus-host disease (GVHD) and clinical responses.

OUTLINE: This is a dose escalation study of bendamustine.

Participants receive rituximab intravenously (IV) over 5-7 hours on days -13 and -6, fludarabine IV over 1 hour and bendamustine IV over 1 hour on days -5 to -3, and tacrolimus IV starting on day -2 and orally (PO) after hospital discharge for 6 to 8 months. Participants with matched unrelated donor (MUD) receive thymoglobulin on days -2 and -1. Participants undergo allogenic stem cell transplant over 30-45 minutes on day 0. Participants receive rituximab IV over 5-7 hours on days 1 and 8 and methotrexate IV over 30 minutes on days 1, 3, and 6. Participants with MUD also receive methotrexate IV on day 11. Participants receive filgrastim (G-CSF) subcutaneously (SC) once daily starting on day 7 until white blood cell counts recover.

After completion of study treatment, participants are followed up every 3 months during year 1 and every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD20 + chronic lymphocytic leukemia (CLL), marginal zone, mantle cell and follicular lymphoma or T-cell lymphoid malignancies who are eligible for allogeneic transplantation.
* Patients with relapsed diffuse large B-cell lymphoma may be included if they were not eligible for autologous transplantation.
* A fully-matched sibling donor or matched unrelated donor.
* Left ventricular ejection fraction (EF) > 40% with no uncontrolled arrhythmias or symptomatic heart disease.
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) > 40%.
* Serum creatinine < 1.6 mg/dL.
* Serum bilirubin < 3 X upper limit of normal.
* Serum glutamate pyruvate transaminase (SGPT) < 3 X upper limit of normal.
* Voluntary signed, written Institutional Review Board (IRB)-approved informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Patient with active central nervous system (CNS) disease.
* Pregnant (positive beta human chorionic gonadotropin [HCG] test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Known infection with human immunodeficiency virus (HIV), human T-lymphotropic virus (HTLV)-I, hepatitis B, or hepatitis C.
* Patients with other malignancies diagnosed within 2 years prior to study day-13 (except skin squamous or basal cell carcinoma).
* Active uncontrolled bacterial, viral or fungal infections.
* History of stroke within 6 months.
* Myocardial infarction within the past 6 months prior to study day 1, or has New York Heart Association (NYHA) class III or IV heart failure or arrhythmias, unstable angina, uncontrolled congestive heart failure or arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiography (ECG) abnormality at screening must be documented by investigator as not medically relevant.
* A prior allogeneic transplant.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has received other investigational drugs within 3 weeks before enrollment.
* Hypersensitivity to bendamustine.
* Prior known refractoriness to bendamustine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bendamustine | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Issa Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Khouri IF, Wei W, Korbling M, Turturro F, Ahmed S, Alousi A, Anderlini P, Ciurea S, Jabbour E, Oran B, Popat UR, Rondon G, Bassett RL Jr, Gulbis A. BFR (bendamustine, fludarabine, and rituximab) allogeneic conditioning for chronic lymphocytic leukemia/lymphoma: reduced myelosuppression and GVHD. Blood. 2014 Oct 2;124(14):2306-12. doi: 10.1182/blood-2014-07-587519. Epub 2014 Aug 21. PMID 25145344
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org